CLINICAL TRIAL: NCT06616181
Title: Effects of Anodal TDCS Applied Over M1 and DLPFC Combined with a Telerehabilitation Exercise Program in Patients with Fibromyalgia: a Randomized Controlled Trial
Brief Title: TDCS and Tele-rehabilitation Exercise in Fibromyalgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Ignacio Hernando Garijo, PhD physiotherapist, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UValladolid02
Record Dates: First submitted 2024-09-22; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Fibromyalgia Syndrome
Keywords: tDCS; exercise; telerehabilitation; home-based exercise; fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Anodal tDCS over M1 + telerehabilitation (Experimental): tDCS over M1: The anode will be placed over the left M1 (C3 according to the International 10-20 system), and the cathode will be positioned over the right supraorbital area (FP2). Once the electrodes are positioned, continuous stimulation at 2mA will be applied for 20 minutes per session, with 30-second initial and final ramp-ups. One session will be administered per week for 12 weeks.
  Telerehabilitation Exercise: Two weekly 50-minute sessions of mixed exercise, including both aerobic and resistance components, will be performed. Aerobic exercises will involve large muscle groups, and resistance exercise will be performed through elastic bands of varying intensity will be used for strengthening exercises. Exercise intensity will be regulated using the modified Borg Rating of Perceived Exertion scale (0-10), with participants maintaining between 4 and 7 points on this scale. The exercises will be monitored through video and weekly phone contact.
  Interventions: Device: Anodal tDCS over M1; Behavioral: Exercise telerehabilitation
- Anodal tDCS over DLPFC + telerehabilitation (Experimental): tDCS over DLPFC: The anode will be placed over the left dorsolateral prefrontal cortex (DLPFC) (F3), and the cathode will be positioned over the contralateral supraorbital area (F8). Once the electrodes are positioned, active tDCS will be applied at 2mA for 20 minutes per session, with 30-second initial and final ramp-ups. One session will be administered per week for 12 weeks.
  Tele-rehabilitation Exercise: Two weekly 50-minute sessions of mixed exercise, including both aerobic and resistance components, will be performed. Aerobic exercises will involve large muscle groups, and resistance exercise will be performed through elastic bands of varying intensity will be used for strengthening exercises. Exercise intensity will be regulated using the modified Borg Rating of Perceived Exertion scale (0-10), with participants maintaining between 4 and 7 points on this scale. The exercises will be monitored through video and weekly phone contact.
  Interventions: Device: Anodal tDCS over DLPFC; Behavioral: Exercise telerehabilitation
- sham-tDCS + telerehabilitation (Placebo Comparator): Sham tDCS: The same electrode placement protocol used for the active tDCS M1 group will be followed in this group. Stimulation will begin with a 30-second ramp-up to reach an intensity of 2 mA, immediately followed by a 30-second ramp-down to 0 mA. This stimulation will be repeated at the beginning and end of the session. Similar to the active tDCS groups, each session will last 20 minutes.
  Telerehabilitation Exercise: Two weekly 50-minute sessions of mixed exercise, including both aerobic and resistance components, will be performed. Aerobic exercises will involve large muscle groups, and resistance exercise will be performed through elastic bands of varying intensity will be used for strengthening exercises. Exercise intensity will be regulated using the modified Borg Rating of Perceived Exertion scale (0-10), with participants maintaining between 4 and 7 points on this scale. The exercises will be monitored through video and weekly phone contact.
  Interventions: Behavioral: Exercise telerehabilitation

INTERVENTIONS:
Device: Anodal tDCS over M1 — The anode will be placed over the left M1 (C3 according to the International 10-20 system), and the cathode will be positioned over the right supraorbital area (FP2). Once the electrodes are positioned, continuous stimulation at 2mA will be applied for 20 minutes per session, with 30-second initial and final ramp-ups. One session will be administered per week for 12 weeks.
  Arms: Anodal tDCS over M1 + telerehabilitation
Device: Anodal tDCS over DLPFC — The anode will be placed over the left dorsolateral prefrontal cortex (DLPFC) (C3 according to the International 10-20 system), and the cathode will be positioned over the right supraorbital area (FP2). Once the electrodes are positioned, continuous stimulation at 2mA will be applied for 20 minutes per session, with 30-second initial and final ramp-ups. One session will be administered per week for 12 weeks.
  Arms: Anodal tDCS over DLPFC + telerehabilitation
Behavioral: Exercise telerehabilitation — Two weekly 50-minute sessions of mixed exercise, including both aerobic and resistance components, will be performed. Aerobic exercises will involve large muscle groups, and resistance training will be performed through elastic bands of varying intensity will be used for strengthening exercises. Exercise intensity will be regulated using the modified Borg Rating of Perceived Exertion scale (0-10), with participants maintaining between 4 and 7 points on this scale. The exercises will be monitored through video and weekly phone contact.

SUMMARY:
This randomized controlled trial aims to analyze the effects of anodal tDCS applied over the primary motor cortex and dorsolateral prefrontal cortex combined with a tele-rehabilitation exercise program in patients with fibromyalgia. The study will compare these effects with each other and with placebo tDCS on the following variables: pain intensity, pain mechanosensitivity, quality of life, fatigue, anxiety, depression, sleep quality, pain catastrophizing, functional capacity, isometric strength, and exercise adherence.

Secondary objectives include:

* Describing the sociodemographic, clinical, and functional characteristics of fibromyalgia patients.
* Comparing exercise intensity levels between patients receiving tDCS on M1, DLPFC, and placebo stimulation.
* Reporting any adverse effects of the intervention. Adult participants with fibromyalgia will be randomized into three groups: a) anodal tDCS over M1 + telerehabilitation, b) anodal tDCS over DLPFC + telerehabilitation, and c) sham-tDCS + telerehabilitation. The intervention will last for 12 weeks. The telerehabilitation exercise program will include an aerobic phase and a resistance phase, with four intensity levels regulated based on the Borg Rating of Perceived Exertion (0-10). The program will be conducted remotely through phone contact, with materials and videos provided to guide exercise execution. tDCS will be applied once per week for 20 minutes at 2 mA, either over M1 or DLPFC.

The dependent variables-pain intensity, fibromyalgia impact, fatigue, anxiety and depression levels, pain catastrophizing, sleep quality, functional capacity, and isometric muscle strength-will be collected in the week prior to the intervention, the week following the intervention, and 12 weeks after its completion. Additionally, pain intensity, fibromyalgia impact, fatigue severity, anxiety and depression levels, pain catastrophizing, and sleep quality will be evaluated during the 6th week of the intervention.

Exercise intensity, exercise adherence, and any adverse effects related to the intervention will be recorded weekly.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 70 years.
* Medical diagnosis of fibromyalgia.Compliance with the latest diagnostic criteria from the American College of Rheumatology.
* Stable medication for at least 12 weeks prior to the start of the study.
* Ability to use communication technologies, such as smartphones and computers.
* Capacity to participate in an aerobic exercise program.
* Access to the internet.
* Proficiency in oral and written Spanish.
* Signed informed consent

Exclusion Criteria:

* Severe psychiatric disorders.
* Uncontrolled cardiovascular, respiratory, metabolic, neurological, rheumatic, or hepatic diseases.
* Concurrent chronic inflammatory or autoimmune disease.
* Contraindications to physical activity.
* Metal implants in the head.
* History of cancer, brain tumor, epileptic episodes, stroke, severe head trauma, or brain surgery.
* Pregnancy or lactation.
* Use of carbamazepine in the past 6 months.
* Changes in medication during the study.
* Participation in other non-pharmacological conservative therapies (e.g., hydrotherapy, electrotherapy, manual therapy, exercise, dry needling) during the study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | At pre-intervention, at weeks 12 and 24.
  Pain intensity will be assessed using the Visual Analog Scale (VAS). Participants will indicate their pain intensity by placing a perpendicular mark on a 100 mm straight line, where the left end represents 'no pain'; and the right end represents 'the worst imaginable pain'. Pain intensity is quantified by measuring the distance in mm from the left end of the line using a ruler.

SECONDARY OUTCOMES:
Pain mechanosensitivity | At pre-intervention, at weeks 12 and 24.
  Pain mechanosensitivity will be assessed by summing the pressure pain thresholds at the 18 tender points described by the ACR in 1990 for the diagnosis of fibromyalgia. The pressure pain threshold is defined as the minimum pressure required to elicit pain. An algometer will be used for measurement. Incremental pressure will be applied at a rate of 1 kg/s at each point until the participant reports the onset of minimal pain. Three measurements will be taken at each point, with a 30-second interval between each. The average of the three measurements will be used to calculate the total sum. The order of measurement for each tender point will be consistent across all participants.
Fatigue | At pre-intervention, at weeks 12 and 24.
  Fatigue will be measured using the Spanish version of the Multidimensional Fatigue Inventory. This scale includes five dimensions: general fatigue, physical fatigue, mental fatigue, reduced activity, and reduced motivation. Each dimension provides a score from 4 to 20, where higher scores indicate greater fatigue.
Sleep Quality | At pre-intervention, at weeks 12 and 24.
  Sleep Quality: Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI). The minimum score is 0 and the maximum is 21 points, with higher scores indicating poorer sleep quality
Pain Catastrophizing | At pre-intervention, at weeks 12 and 24.
  Pain Catastrophizing: Pain catastrophizing will be assessed using the Spanish version of the Pain Catastrophizing Scale. It has a minimum score of 0 and a maximum score of 52 points, with higher scores indicating greater catastrophizing thoughts about pain.
Isometric Strength | At pre-intervention, at weeks 12 and 24.
  Maximum isometric muscle strength will be measured for elbow flexors and knee extensors by hand-held dynamometry.
Exercise Adherence | At weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12.
  Exercise adherence will be estimated as the percentage of completed sessions out of the 24 scheduled sessions. This will be tracked weekly using Google Forms to record the number of sessions completed.
6-Minute Walk Test | At pre-intervention, at 12 and 24 weeks.
  In this test, the distance in meters that the participant can walk at a fast but comfortable pace, without running, within 6 minutes will be measured. Two cones will be placed 20 meters apart in an unobstructed hallway.
30-second Chair Stand Test | At pre-intervention, at weeks 12 and 24.
  This test consists of measuring the number of times the participant can stand up and sit down again in a chair without armrests within 30 seconds.
Fibromyalgia Impact | At pre-intervention, at weeks 12 and 24.
  Fibromyalgia Impact: The impact of fibromyalgia will be measured using the Spanish version of the Revised Fibromyalgia Impact Questionnaire (FIQ-R). The scale ranges from 0 to 100 points, where higher scores indicate a greater impact of fibromyalgia.

OTHER OUTCOMES:
Exercise intensity | At weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12.
  Exercise intensity will be recorded after each session by Google Forms.
Adverse events | At weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12.
  Adverse events will be recorded after each session through Google Forms.

IPD SHARING:
Plan to Share IPD: No